CLINICAL TRIAL: NCT05770635
Title: A Prospective, Multicenter, Randomized Controlled Trial to Evaluate the Safety and Efficacy of Polyvinyl Alcohol Embolization Microspheres for Transarterial Chemoembolization of Primary Liver Cancer
Brief Title: Polyvinyl Alcohol Embolization Microspheres
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Huihe Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSP-V-01
Record Dates: First submitted 2023-03-05; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyvinyl alcohol embolization microspheres (Huihe Medical) and chemotherapy drug (Experimental): The experimental group received chemotherapy drug + polyvinyl alcohol embolized microspheres (Huihe Medical) for target lesion TACE (Trans-Arterial Chemoembolization)treatment.Experimental group and control group were selected to use iodide oil according to the condition of subjects.
  Interventions: Device: Polyvinyl alcohol embolization microspheres (Huihe Medical) and chemotherapy drug
- Embosphere and chemotherapy drug (Other)
  Interventions: Device: Embosphere and chemotherapy drug

INTERVENTIONS:
Device: Embosphere and chemotherapy drug — chemotherapeutic drug + embolic Embosphere;Iodide is selected according to the subject's condition
  Arms: Embosphere and chemotherapy drug
Device: Polyvinyl alcohol embolization microspheres (Huihe Medical) and chemotherapy drug — chemotherapy drug+Polyvinyl alcohol embolization microspheres (Huihe Medical);Iodide is selected according to the subject's condition
  Arms: Polyvinyl alcohol embolization microspheres (Huihe Medical) and chemotherapy drug

SUMMARY:
To evaluate the safety and efficacy of polyvinyl alcohol embolization microspheres developed and manufactured by Shanghai Huihe Medical Technology Co., LTD. (hereinafter referred to as Huihe Medical) for transarterial chemoembolization of primary liver cancer using a prospective, multi-center, randomized controlled method

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old; age ≤85 years old; regardless of gender
2. Patients with CNLC Ib, IIa, IIb, IIIa who need transarterial chemoembolization (TACE) therapy and are not suitable for or refuse surgical resection, liver transplantation, and ablation, and patients with stage IIIb primary liver cancer who are expected to benefit from TACE therapy to control the growth of intrahepatic tumors;
3. Child-Pugh A or B (less than 10 points);
4. performance status (PS) score of ECOG 0~2;
5. The patient had at least one measurable tumor lesion without embolization (maximum diameter of the target lesion ≤10cm);
6. Those who agree to participate in the clinical trial and voluntarily sign the informed consent;

Exclusion Criteria:

1. Patients whose target lesions had received embolization therapy, whose target lesions had received other local treatments besides TACE (including but not limited to surgery, radiotherapy, hepatic arterial perfusion, radiofrequency ablation, cryoablation or percutaneous ethanol injection) within 1 month, or who had received first TACE therapy for target lesions combined with ablation/radiotherapy after inclusion;
2. The proportion of tumor in total liver volume was ≥70%;
3. Patients with distant extensive metastasis or other malignant tumors;
4. The expected survival time is less than 3 months;
5. Cachexia or multiple organ failure;
6. Severe liver dysfunction (Child-Pugh grade C), including jaundice, hepatic encephalopathy, refractory ascites, or hepatorenal syndrome;
7. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 times the upper limit of normal or >250U/L, and ≥2 times the upper limit of normal after 1 week of liver protection and antiviral treatment;
8. Renal dysfunction: patients with serum creatinine > 2mg/dL;
9. Blood leukocytes and platelets decreased significantly, leukocytes < 3.0×109/L, platelets < 50×109/L (except patients with hyperplenism and chemotherapy myelosuppression);
10. Bleeding and thrombotic tendency: patients with known hereditary or acquired bleeding and thrombotic tendency (e.g., hemophiliacs, uncorrectable coagulation disorders, thrombocytopenia, hyperplenism, etc.), active peptic ulcer or gastrointestinal bleeding within 30 days; Arteriovenous thrombosis occurred in the past 6 months (until enrollment);
11. Patients with active hepatitis or severe infection who cannot be treated with TACE simultaneously;
12. Patients with complete obstruction of the main portal vein and unable to restore portal blood flow through compensatory collateral branches of the portal vein;
13. The target focal blood supply arteries cannot be treated with TACE or have the risk of embolization (vascular access endangers normal areas, arteriovenous fistula, portal fistula, etc.);
14. Subjects who predicted that the target lesion would require more than three TAces; Uncontrolled diabetes mellitus; 15.

16. People with known severe allergy to contrast agents, iodine contrast agents or embolic materials; 17. Pregnant/lactating women, or those who plan to give birth; 18. Patients who are participating in clinical trials of other drugs or devices and have not been in the group or have been in the group for less than 1 month; 19. Persons without the ability to make independent decisions or with mental illness; 20. Other patients deemed unsuitable for this clinical trial by the investigator;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2024-12-28 (Estimated); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) 1 month after the last TACE -mRECIST evaluation | 1 month after the last TACE -mRECIST evaluation
  Target lesions of subjects were treated with TACE for 1-3 times as needed, and the last evaluation of target lesions before enrollment was used as baseline tumor evaluation. One month after the last TACE, all subjects underwent plain CT and enhanced MRI examinations, which were compared with the baseline of target lesions. The efficacy was evaluated according to the mRECIST (Modified Response Evaluation Criteria in Solid Tumors)for the treatment of solid tumors in target foci. For example, multiple tumor foci were embolized at the same time, and the two largest target foci were selected as the evaluation foci:

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Huihe Healthcare Tecnology Co.,Ltd., Shanghai, Shanghai Municipality, China